CLINICAL TRIAL: NCT01882894
Title: Efficacy of a Custom Temporary Foot Orthosis for Plantar Fasciitis Treatment: A Randomized Controlled Trial.
Brief Title: Efficacy of a Custom Temporary Foot Orthosis for Plantar Fasciitis Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Puget Sound (Other)
Responsible Party: Principal Investigator, Robert Boyles, Clinical Associate Professor, University of Puget Sound
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PFO Trial
Record Dates: First submitted 2013-06-17; First posted 2013-06-21 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Plantar Fasciitis
Keywords: Plantar fasciitis, orthotic, functional outcome
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Custom PFO orthosis (Experimental): This is a custom made orthosis
  Interventions: Device: Custom PFO
- Faux foot orthosis (Placebo Comparator): Foam insert without arch support
  Interventions: Other: Faux orthosis

INTERVENTIONS:
Device: Custom PFO — PFO made out of thermoplastic material molded to the patient's foot
  Arms: Custom PFO orthosis
Other: Faux orthosis — Foam cut out
  Arms: Faux foot orthosis

SUMMARY:
The aim of this randomized control trial is to identify the possible effectiveness of the temporary use of an inexpensive, custom-made plantar fascia orthotic (PFO).

DETAILED DESCRIPTION:
A. Background Plantar fasciitis is the most common foot complaint in America, affecting approximately 10% of people during their life time.9 It can be a painful and debilitating condition which appears in both sedentary and active populations. A survey performed by the Foot and Ankle Special Interest Group of the Orthopedic Section, APTA, found that 100% of therapists reported PF as the most common foot condition seen in their clinic. 9 Approximately one million patients visit physicians for the diagnosis and treatment of plantar fasciitis.10 Chronic plantar fasciitis, previously thought to be an inflammatory condition caused by repetitive microtearing of the plantar fascia, is now thought to be a degenerative condition.5 The plantar aponeurosis, or fascia, functions to provide static support of the longitudinal arch and dynamic shock absorption. It consists of 3 bands: lateral, medial, and central. The central band originates from the medial tubercle of the calcaneus and travels across the metatarsal heads to the phalanx of each toe.9 In the acute stage, pain is commonly localized to the origin of the medial and central bands at the plantar surface of the calcaneus.6 This pain is usually classified as a sharp or knife-like pain upon initial standing. The pain occurs after a period of non-weight bearing and is often the worst in the morning. Those in the chronic stages may report pain as being dull and achy. Pain in this stage may also extend beyond the medial tubercle, extending into the central and lateral bands. Pain at this stage does not usually subside after a few minutes of walking as seen in the acute phase.6 Many factors contribute to the development of plantar fasciitis. Anatomy, biomechanics and environment are factors which contribute to the development of this condition.6 Pes planus, pes cavus feet, limited dorsiflexion, tight Achilles tendon, tight hamstrings and obesity fall beneath anatomical causations. Biomechanical factors include weak plantar flexor muscles and excessive subtalar joint pronation. Environmental factors include weight bearing activities, foot wear and trauma.6 Certain diseases also place an individual at increased risk. These may include diabetes, peripheral vascular neuropathy, Paget's disease, Reiter's syndrome, and other autoimmune and neurologic disorders.8 Diagnosis is mostly made upon clinical assessment and findings for classifying a patient with heel pain into the International Statistical Classification of Diseases and Related Health Problems category of plantar fasciitis and associated International Classification of Functioning Disability and Health impairment based category of heel pain.9 To date, there is no specific treatment of choice for patients with plantar fasciitis. Multiple studies have been conducted on various conservative treatment techniques but according to Crawford et al's Cochrane Review, "There is limited evidence upon which to base clinical practice." 1 The options include: modalities, manual therapy, stretching, taping, night splints, steroid injections and orthotic devices. Of all the previous interventions, there is strong evidence to support the use of orthotic devices to provide temporary relief of symptoms.9 Traditional orthotic devices are designed and casted with the subtalar and midtarsal joints in a neutral position. They are hypothesized to limit excessive pronation, optimize biomechanical loading of the foot, and off load the plantar fascia.10 Additionally, custom orthotics are costly and may require the specialty services of an orthotist to cast the individual. Despite the cost and time-intensive manufacturing process, custom orthotics are often worn for life and may prove to be ineffective after 3 months.9 A recent pilot study proposed the benefit of temporary foot orthoses casted in equinos position for plantar fasciitis treatment.2,3 As opposed to the traditional casting method of subtalar and midtarsal joints in neutral, the equinos position places the patient's foot in full plantar flexion and inversion. This casting position is hypothesized to put the plantar fascia in a slackened position, therefore reducing weight-bearing on the damaged tissue.2 Consequently, the aim of this randomized control trial is to identify the possible effectiveness of the temporary use of an inexpensive custom-made plantar fascia orthotic (PFO), fabricated in equinos position of the foot.

B. Project Description Prior to study commencement a training session will be provided to educate and ensure all investigators are able to perform examination, casting and accurately provide instruction to all participants. All investigators will also be trained in distribution and analysis of all outcome measures to be used in the study.

The study will begin with subjects completing a medical screening questionnaire. All subjects will then go through a formal physical examination that is conducted by one of the investigators. Subjects meeting the criteria for admission and consenting to participate in the study, will sign an informed consent form, and be included in the study. Subjects will be assigned to a control or experimental group via a random number generator. Subjects will then complete two outcome measures to collect baseline data, the Foot and Ankle Ability Measure (FAAM) and a Numeric Pain Rating Scale (NPRS). The FAAM has been shown to be a valid and reliable self-reported outcome measure of lower leg, ankle, and foot function of a range of musculoskeletal disorders in a physical therapy setting. The FAAM asks patients to rate level of difficulty in several activities of daily living and in sport specific activities. The NPRS asks patients to rate the intensity of first step heel pain on scale of 0-10, with 0 equal to no pain and 10 equal to worst pain ever experienced. Additionally, a GRC has been shown to be a valid and reliable method of assessing changes in quality of life over time. A Global Rating of Change (GRC) will be collected throughout the study (baseline, two weeks, four weeks, twelve weeks, and six months). Upon initial evaluation, researchers will also complete a Foot Posture Index (FPI-6) for each subject to classify static foot posture in a standing position. The FPI-6 looks at multiple bony landmarks of the foot in a full weight-bearing position and gives each landmark a score based on its position during standing. A total score is produced to describe the patient's foot type.

Following collection of baseline data, one of the researchers will begin fabricating the individuals in the experimental group for a custom-made PFO. The custom-made PFO will be completed by placing subject's foot in the equinos (plantar flexed and inverted) position. The custom-made PFO will be created from Aqua-Plast casting material. After heating the Aqua-Plast material, researchers will drape the material over their forearm to ensure that it isn't too hot for the subject. When the orthosis is hardened, the subject will place it in his/her shoe (after removing any shoe liners). Researchers will trim, stretch, or pad the orthosis as needed to make sure it is completely comfortable. If the orthosis is rubbing or is otherwise found to be uncomfortable, the rough edges will be reheated and smoothed with a finger or a grinder will be used to taper the edges. Subjects will be told to come in at any time to make any needed changes. Full instructions for construction of the custom-made PFO will be included.

Control group subjects will be asked to wear a faux orthotic that will be constructed of a soft material that will cushion, but not support, the plantar fascia. Subjects will be asked to wear either the PFO or faux orthotic at all times while weight bearing for a two week time frame during the initial treatment period. An exception will be made for showering, in which the subjects will be instructed to weight-bear on the lateral side of the foot to avoid pronation and pulling on the plantar fascia. After two weeks, subjects will be weaned off of the orthotic for one week. Weaning includes wearing orthotic 8 hours per day, following a stretching program that includes a Windlass (plantar fascia) stretch with soft tissue mobilization and calf stretch, and ankle range of motion exercises.

The plantar fascia stretch will consist of the patient sitting and placing his/her affected foot crossed over the opposite knee and then using his/her hand to pull the toes and ankle back towards the anterior surface of the lower leg. Once in position the patient will continue to hold the stretch and apply deep pressure to the plantar fascia from heel to toe with his/her fingers, thumbs, or knuckles. This activity will be carried out for three minutes.2 For the gastrocnemius and soleus stretch, the patient will stand 46-61cm away from a wall, place his/her hands on the wall at shoulder level, and then bend the knee of the uninvolved leg, while extending the leg of the involved side so that the foot is about 30cm back. Keeping the back knee straight, the patient will lean slowly in to the wall while maintaining his/her heel on the floor and hold this stretch for 30 seconds. This stretch will be repeated four times per session.

Ankle range of motion exercises will be completed prior to the patient getting out of bed each morning and will consist of the patient: dorsiflexing and plantar flexing his/her ankle on the involved side, with the knee straight and with the knee bent, ten times in each position; and performing clockwise and counter-clockwise ankle circles ten times in each direction.

Participant's outcome indicators will be recorded at the end of two weeks, four weeks, twelve weeks, and six months following casting. The following outcome measures will be used: NPRS, FAAM, FPI-6, and GRC. Subjects will be seen in the clinic for the initial exam, two, four, and twelve week follow-up intervals, with the final six month follow-up conducted via e-mail, telephone, and postal mail, per the subject's preference.

C. Subject Recruitment Convenience sampling will be implemented in selecting up to 60 subjects from a population of individuals with chronic plantar fasciitis who have either received, or not received treatment in the previous three months for the same condition. Following IRB approval, clinical sites, running stores and university campus will be solicited for recruitment of participants. Inclusion for our sample will include: age 18 years or older, able to tolerate the physical examination and treatment procedures, symptoms greater than four weeks, able to read, write, and speak sufficient English to be able to complete the outcome tools, plus two of three of the following: symptom reproduction with palpation of the proximal plantar fascia insertion and/or mid substance of plantar fascia, positive Windlass test and/or first step pain after period of inactivity. A positive Windlass test consists of symptom reproduction when the first metatarsophalangeal joint is placed into passive extension while the patient is in a standing position. Exclusion criteria for our sample will include: current symptoms consistent with a lumbar radiculitis, radiculopathy, or myelopathy, history of foot or ankle fracture with or without the presence of hardware from an open reduction internal fixation, positive tarsal tunnel syndrome test, known or suspected pregnancy, and systemic Rheumatic disease, or those undergoing litigation for any medical condition.

D. Confidentiality of Data The subjects will be carefully screened so as to eliminate any possible risks from the protocol. The screening, evaluation and treatment will be performed by physical therapists or senior physical therapy students fully trained to perform all procedures under their scope of practice. As is the standard of practice, the investigator will communicate with the subject during the entire process to ensure that each subject is informed throughout the treatment protocol. All records will be kept confidential per HIPAA and university operating procedures. No personal identifying information about any subject in the study will be released to anyone. Data will be secured in locked rooms and on computers that are password-protected and only accessible to the investigators in the study. In the unlikely event of an adverse response to treatment, subjects will be provided appropriate physical therapy and medical intervention.

E. Risk to Subjects The effect of custom-made orthotics fabricated with Aquaplast for the treatment of plantar fasciitis is not well documented in the literature. However, this is a non-invasive, patient-directed treatment with minimal known risks, and considered safe and ethical practice. A faux orthotic is also a low-risk treatment method that does not pose any risk to the health of control subjects. Risks would include blisters and abrasions from the orthotic rubbing on the foot and soreness or pain associated with the changes of joint alignments due to the orthotic. The subjects will be instructed to return immediately, or call the researchers, if there is any pain associated with the wear of either orthotic.

F. Benefits Experimental participants will benefit from this study by receiving treatment that will attempt to eliminate, or significantly reduce, heel pain associated with plantar fasciitis, which may yield an effective, non-invasive, treatment strategy to eliminate the symptoms associated with plantar fasciitis. Upon completion of the study subjects in the control group will be offered the PFO, if results show significant improvement for the experimental group. All subjects in the experimental group will be able to keep their PFO's.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able to tolerate the physical examination and treatment procedures, have symptoms greater than four weeks, able to read, write, and speak sufficient English to be able to complete the outcome tools, plus two of three of the following: symptom reproduction with palpation of the proximal plantar fascia insertion and/or mid substance of plantar fascia, positive Windlass test and/or first step pain after period of inactivity

Exclusion Criteria:

* current symptoms consistent with a lumbar radiculitis, radiculopathy, or myelopathy, history of foot or ankle fracture with or without the presence of hardware from an open reduction internal fixation, positive tarsal tunnel syndrome test, known or suspected pregnancy, and systemic Rheumatic disease, or those undergoing litigation for any medical condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-04 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Foot Ankle Ability Measure (FAAM) to measure change from Baseline at 4 time frames | Baseline, 2wks, 4 wks, 12 wks, 6 months
  The FAAM has been shown to be a valid and reliable self-reported outcome measure of lower leg, ankle, and foot function of a range of musculoskeletal disorders in a physical therapy setting

SECONDARY OUTCOMES:
Global Rating of Change (GRC) to measure perceived change at 4 follow-up periods | 2 wks, 4 wks, 12 weeks, 6 months
  The GRC is a 15 point scale used to measure patient's perceived change in their health status compared to baseline.

OTHER OUTCOMES:
Numeric Pain Rating Scale (NPRS) to measure change from baseline at 4 different time frames | Baseline, 2 wks, 4 wks, 12 wks and 6 months
  THe NPRS is a 11 point self report measure for rating the patient's pain. Will will be using the NPRS to rate first step pain.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Puget Sound, Tacoma, Washington, United States